CLINICAL TRIAL: NCT03074019
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Pilot Study on the Effect of a Novel Prebiotic, XOS95, on the Human Gut Microbiome
Brief Title: Pilot Study on the Effect of a XOS95 on the Human Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prenexus Health (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRENRPD-150002-RPD01
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Healthy
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, 3-arm, parallel, dose ranging study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Xylooligosaccharide (Low Dose) (Experimental): 1.5g XOS95 + 1.5g Maltodextrin powder, taken orally mixed in water, once daily
  Interventions: Dietary Supplement: Xylooligosaccacharide
- Xylooligosaccharide (High Dose) (Experimental): 3g XOS95 powder, taken orally mixed in water, once daily
  Interventions: Dietary Supplement: Xylooligosaccacharide
- Placebo (Placebo Comparator): 3g maltodextrin powder, taken orally mixed in water, once daily
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Xylooligosaccacharide — XOS95 powder
  Other Names: XOS95
  Arms: Xylooligosaccharide (High Dose); Xylooligosaccharide (Low Dose)
Dietary Supplement: Maltodextrin — Maltodextrin powder
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to assess the efficacy of a novel prebiotic, XOS95, at two different dosages, in comparison to a placebo by assessing shifts in microbial populations after 8 weeks of supplementation, assessed as changes in abundance of microbial populations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 18 - 60 (inclusive)
* Healthy as determined from medical history
* Non-smoker, or ex-smoker ≥6 months
* Body mass index 18.5 - 27.5kg/m2 (inclusive)
* Female subjects of childbearing potential [i.e. not surgically sterilized or post-menopausal (greater than one year since last menses)] must have negative urine pregnancy test and must be using an effective birth control method , defined as:

  * Continuous use of oral or long acting injected contraceptive for at least 2 months prior to study entry , or
  * Use of an intra-uterine device or implantable contraceptive, or
  * Use of double barrier methods of birth control, or
  * Abstinence from heterosexual intercourse
* Willing to avoid alcohol consumption for 24 h prior to every clinic visit
* Willing to maintain their regimens of medications and supplements known to alter GI function (including, but not limited to, iron supplements, calcium, and anti-depressants)
* Willing to maintain a stable body weight, activity level and dietary pattern except for use of the study products, as directed
* Willing and able to provide informed written consent

Exclusion Criteria:

* Pregnancy or lactation, or subject unwilling to take appropriate contraceptives for the duration of the study
* Use of prescription non-steroidal anti-inflammatory drugs (or daily use of over the counter non-steroidal anti-inflammatory drugs >1month), steroids, corticosteroids, or any other prescription anti-inflammatory drugs within 3 months prior to visit 1
* Individuals taking any over the counter or prescription medications, including natural health products, that may alter lipid profiles including, but not limited to fish oil (omega-3 fatty acids), statins, fibrates, bile acid exchanger resin, phytosterols, niacin or its analogues, carnitine, polyglucosamines (Chitosan) or other lipid-binding ingredients within the 3 months prior to visit 1
* Individuals taking any over the counter or prescription medications, including natural health products that may alter blood glucose (e.g. biguanides (Metformin), Alpha-lipoic Acid (ALA), Gymnema sylvestre) or insulin modulating medications (e.g. sulfonylureas, meglitinides, D-phenylalanine derivatives, thiazolidinediones, DPP-4 inhibitors, alpha-glucosidase inhibitors, bile acid sequestrants within 3 months prior to visit 1
* Use of proton pump inhibitors or medications which inhibit peristaltic movement (e.g. opioids, loperamide)
* Unstable use (i.e. initiation or change in dose) of antihypertensive medications or thyroid hormone replacement medications within 3 months prior to visit 1
* Use of any weight-loss programs or weight-loss medications (prescription or over-the counter) including, but not limited to, lipase inhibitors, within 3 months prior to visit
* Use of over the counter or prescription laxatives or stool softeners within 1 month prior to baseline (V2)
* Use of antibiotics (other than topical) within 2 months prior to baseline (V2)
* Use of prebiotic or fiber supplements (e.g. fructans and galacto-oligosaccharides (FOS, GOS), psyllium, fiber, inulin, glucomannan, acacia fiber/gum) or probiotic supplements (i.e. live microorganisms) within 4 weeks of baseline (V2)
* Consumption of specific functional prebiotic- or probiotic-rich foods within 4 weeks of baseline (V2) (Appendix 3)
* History of blood clotting disorders or use of coagulation-inhibiting drugs (e.g. warfarin)
* Individuals with achlorhydria
* Presence of major diseases such as diabetes, gastrointestinal, endocrine, cardiovascular, pancreatic, renal, or liver disease
* Chronic diarrhea or constipation, irritable bowel syndrome, celiac disease, gluten-sensitive enteropathy, or inflammatory bowel disease
* Abdominal or gastrointestinal surgery within the previous 12 months or planned abdominal or gastrointestinal surgery or procedures such as colonoscopy in the next 4 months
* Recent gastrointestinal food-borne illness (within 1 month prior to visit 1)
* History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.)
* History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in the past 5 years
* Uncontrolled hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
* Abnormal laboratory test results of clinical significance, including, but not limited to ALT or AST ≥1.5X the upper limit of normal at screening (visit 1)
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day
* Extreme dietary habits (e.g. vegan or very low carbohydrate diets, gluten-free diet, low FODMAP diet)
* Subject has a known allergy or intolerance to the test products or placebo
* Subject is unwilling or unable to abide by the requirements of the protocol
* Any condition that would interfere with the subject's ability to comply with study instructions, might confound the interpretation of the study, or put the subject at risk
* Subject has taken an investigational health product or has participated in a research study within 30 days prior to first study visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Effect of XOS95 on abundance of microbial populations by 16S RNA sequencing of feces | 8 weeks

SECONDARY OUTCOMES:
Effect of XOS95 on short chain fatty acid production measured in the feces | 8 weeks
Effect of XOS95 on gastrointestinal bacterial counts in the feces | 8 weeks
Effect of XOS95 on fasting blood glucose | 4 and 8 weeks
Effect of XOS 95 on post-prandial glucose response | 8 weeks
  2 hour post-prandial response to a 75g oral glucose challenge
Effect of XOS 95 on lipid profile parameters | 4 and 8 weeks
  Effect of XOS 95 on lipid profile parameters (Total cholesterol, LDL-C, HDL-C and triglycerides)
Effect of XOS 95 on C-reactive protein | 8 weeks
Effect of XOS on abdominal discomfort assessed by daily questionnaire | 4 and 8 weeks
Effect of XOS on general well-being assessed by daily questionnaire | 4 and 8 weeks
Effect of XOS on total Gastrointestinal Quality of Life Index (GIQLI) scores | 4 and 8 weeks

OTHER OUTCOMES:
Adverse events | 8 weeks
  Number of subjects with a treatment emergent adverse effect

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrasource Diagnostics Inc., Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No